CLINICAL TRIAL: NCT02305225
Title: Cortical Excitability and Decision Making After Total Sleep Deprivation and Sleep Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Baumann (Other)
Responsible Party: Sponsor-Investigator, Christian Baumann, Associate professor and leading physician, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-0496
Record Dates: First submitted 2014-11-07; First posted 2014-12-02 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Acute and Partial Sleep Deprivation

ARMS (2):
- SDSR (Experimental): first total then partial Sleep deprivation
  Interventions: Behavioral: Sleep Deprivation
- SRSD (Experimental): first partial then total Sleep deprivation
  Interventions: Behavioral: Sleep Deprivation

INTERVENTIONS:
Behavioral: Sleep Deprivation

SUMMARY:
The investigators examine changes in decision making, vigilance and cortical excitability in healthy male subjects undergoing total acute sleep deprivation (40 hours) on the one hand, and chronic partial sleep restriction (7 nights with 5 instead of 8 hours in bed per night) on the other hand, in a cross over controlled manner. The investigators hypothesize that total sleep deprivation, as well as partial sleep restriction lead to impairments in decision making and vigilance, and enhanced cortical excitability.

Beside these three primary outcomes, the investigators also assess changes in sleep by EEG, dim light melatonin onset, skin temperature, subjective mood and sleepiness, working memory, and also collect saliva samples.

ELIGIBILITY:
Inclusion Criteria:

* Male (in female subjects, menstrual cycle influences sleep)
* Age between 18-35 years
* Right-handedness
* Good general health
* Signed Informed Consent after being informed

Exclusion Criteria:

* Contraindications on ethical grounds
* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc)
* Known or suspected non-compliance, drug or alcohol abuse (> 5dl wine/ >1l beer daily)
* Regular medication intake
* Enrolment into a clinical trial within last 4 weeks
* History of seizure or a family history of epilepsy
* Diseases or lesions of the nervous system (acute or residual included neurological and psychiatric diseases)
* History of any moderate or heavy head trauma
* Sleep disorders (e.g. Insomnia, sleep apnea, restless leg syndrome, narcolepsy, etc.)
* Sleep complaints in general or EDS
* Irregular sleep-wake rhythm (e.g. shift working)
* Long (> 9 hours per night) or short sleepers (< 7hours per night)
* Sleep efficiency ≤ 80%
* Travelling with time lag less than 1 month ago (or planning to do so within 1 month prior to the study)
* Body Mass Index < 19 or > 30 kg/m2

  * 5 drinks or food items containing caffeine per day
  * 10 cigarettes per day
* Student of one of the following subjects: Mathematics, Physics, Computer Science, Economics, or Psychology (since students of these subjects have profound knowledge of probability calculations, which could interfere with our measurements in decision making)
* The following additional exclusion criteria apply only to subjects with TMS sessions
* History of frequent and/or heavy headache respectively migraine
* History of claustrophobia
* Hearing disorder
* Magnetic Resonance Imaging (MRI) contraindication (such as pacemaker implanted pumps, shrapnel, etc.; full MRI screening form will be filled out - see -Entrance questionnaires)
* No clear TMS evoked potential in the target area during the screening assessment
* These subjects will be invited to participate in the study with no TMS sessions, the other protocol being identical

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Change in cortical excitability after Chronic Sleep Deprivation as measured by TMS evoked responses in the EEG | Change from Baseline to after 7 nights of chronic Sleep Deprivation
  amount of activation in the electroencephalography (EEG) evoked by single-pulse transcranial magnetic stimulation (TMS)
Change in Reaction Times after Chronic Sleep Deprivation as measured by the Psychomotor Vigilance Task | Change from Baseline to after 7 nights of chronic Sleep Deprivation
  Reaction times in the Psychomotor vigilance task
Change in risk taking and financial impulsivity as measured by the Amount of risky options chosen in the risk task and the amount of financial impulsive choices in the Delay Discount Task | Change from Baseline to after 7 nights of chronic Sleep Deprivation
  Risk Task (adapted from Levy et al.) Delay Discounting Task (Kirby et al.)

SECONDARY OUTCOMES:
Slow Wave Activity during Sleep as measured by the power in the EEG in the frequency range of 1-4.5 Hz | Baseline, 1st Recovery Night of total Sleep Deprivation, 5th, 6th, 7th night of partial Sleep Deprivation, 1st Recovery Night from partial Sleep Deprivation
  Slow wave activity recorded during the night in the electroencephalography
Dim Light Melatonin Onset as measured by the melatonin concentration in hourly collected saliva samples | Baseline, 1st evening after partial Sleep Deprivation, 7th to 14th evening after partial Sleep Deprivation
  Melatonin concentration curve in saliva samples collected hourly prior to going to bed
Skin Temperature profiles as measured by skin temperature sensors (Celsius) | from 1 week prior to partial Sleep Deprivation to 8-14 days after
  Skin temperature (Celsius) is measured every 5 minutes
Mood ratings as measured by a visual analog scale | 2 Baseline Days (prior to both parts), 1st Day of total Sleep Deprivation, 1st Day of Recovery from total Sleep Deprivation, 6th, 7th & 8th Day of partial Sleep Deprivation, 8th to 14th Day of Recovery from partial Sleep Deprivation
  Mood Ratings from 1-10
subjective sleepines as measured by the stanford sleepiness scale | 2 Baseline Days (prior to both parts), 1st Day of total Sleep Deprivation, 1st Day of Recovery from total Sleep Deprivation, 6th, 7th & 8th Day of partial Sleep Deprivation, 8th to 14th Day of Recovery from partial Sleep Deprivation
  Stanford sleepiness scale
Working Memory performance as measured by errors of comission and omission the n-back Task | 2 Baseline Days (prior to both parts), 1st Day of total Sleep Deprivation, 1st Day of Recovery from total Sleep Deprivation, 6th, 7th & 8th Day of partial Sleep Deprivation, 8th to 14th Day of Recovery from partial Sleep Deprivation
  2-back and 3-back task: measures of comission and omission
metabolic profile as measured by metabolites in saliva | Baseline Day 1, 1st Day of total Sleep Deprivation, 8th Day of partial Sleep Deprivation
  Screening for metabolites that are changes due to sleep loss

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland